CLINICAL TRIAL: NCT00310687
Title: A Phase IV, Single Centre, Open-label Study to Evaluate the Persistence of Antibodies in Adolescents 14-16 Years of Age, Vaccinated With Chiron Meningococcal C Conjugate Vaccine During the 1999-2001 UK MenCC Immunization Campaign, at One Year After Either a Challenge Dose of Aventis Pasteur MSD Meningococcal A/C Polysaccharide Vaccine or a Booster Dose of MenC Vaccine, in Parallel to Subjects Aged 11-20 Evaluated at 4 Years After Vaccination During the 1999-2001 UK MenCC Immunization Campaign
Brief Title: Persistence of Immune Response After Vaccination With MCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M14P2E1; Impact N° 919
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prevention of Meningococcal Infection
Keywords: Prevention of Meningococcal Meningitis; vaccines; conjugate; immunology; antibody persistence
MeSH Terms: interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: BLOOD DRAW

SUMMARY:
Persistence of Immune response after vaccination with MCC

ELIGIBILITY:
Inclusion Criteria:

* healthy adolescents vaccinated with Meningococcal C Conjugate vaccine

Exclusion Criteria:

* ascertained or suspected disease caused by N. meningitidis
* household contact with individuals with proven N. meningitidis serogroup C infection
* significant acute or chronic infections
* any other serious disease

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1244
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
persistence of memory response to N. meningitidis serogroup C as measured by serum bactericidal activity at one year after either a challenge with 1/5 of a dose of Meningococcal A/C Polysaccharide vaccine or a booster dose of MenC Vaccine.

SECONDARY OUTCOMES:
Evaluation and comparison of the persistence of antibodies against N. meningitidis serogroup C as measured by hBCA
Evaluation of the immunological response (ELISA) to N. meningitidis serogroup C

CONTACTS AND LOCATIONS:
Overall Officials: Vaccines - Information Services, Principal Investigator — Novartis Vaccines & Diagnostics
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Headington, Oxfordshire, United Kingdom